CLINICAL TRIAL: NCT04010981
Title: Comparison of the Effectiveness of Virtual Reality and Video Assisted Exercises in Pediatric Chronic Kidney Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Irmak ÇAVUŞOĞLU, Principal Investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.30224
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Kidney Disease; Physical Activity; Exercise Addiction
Keywords: Pediatric Chronic Kidney Disease,; virtual reality; physical therapy; exercise; Nintendo wii; Video based exercise
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study grup-Virtual reality- Nintendo Wii Fit exercise group (Experimental): in this group patients will complete 12 sessions of virtual reality exercise - Nintendo Wii Fit Plus, 30-minute training sessions with strengthening exercises for the lower extremities and upper extremities, aerobic and balance exercises, two days a week. They will do 5 minute warm-up exercises before stretching, stretching exercises and 5 minute cooling exercises at the end of the session, as well as breathing exercises and will attend a total of 50 minutes of treatment.
  Interventions: Other: study group
- control group-home based video exercise group (Active Comparator): Patients will be join home based exercises two days a week during 12 sessions .we will prepare for the lower and upper extremity features similar to Nintendo Wii Fit exercises 30 minutes of video game exercise practices, 5 minutes warm-up exercises, 5 minutes cooling exercises and complete the 50-minute training session with the breathing exercises we will teach them. In addition to exercise sessions, patients will record their activities (walking, cycling, swimming ına) in daily life schedules with their pedometers. Thus, changes in physical activity levels will be monitored.
  Interventions: Other: control group

INTERVENTIONS:
Other: study group — The treatment protocol will consist of Nintendo wii fit virtual reality exercises (yoga,aerobic exercises,muscle strengthening exercises)
  Other Names: virtual reality based therapy -aerobic exercises, stretching exercises
  Arms: study grup-Virtual reality- Nintendo Wii Fit exercise group
Other: control group — The treatment protocol will consist of home based video exercises ;yoga,aerobic exercises,muscle strengthening exercises
  Other Names: home based video exercise group
  Arms: control group-home based video exercise group

SUMMARY:
In this study, we aim to improve respiratory function and balance of decreased muscle strength, decrease fatigue values, improve quality of life, improve inflammation findings and GFR ( Glomerular filtration rate) values in pediatric chronic kidney patients with virtual reality exercise applications.

DETAILED DESCRIPTION:
1.Group - Working group: Virtual reality technology (Nintendo Wii Fit Plus) exercise group 2.Group-Control group: home-based video games will be divided into groups that exercise.

Measurements of functional capacity, muscle strength, quality of life, depression, fatigue and physical activity levels, medical values (pulmonary function test values, inflammation level values, glomerular filtration rate level values) of both groups will be recorded before and after treatment.

In the study group treatment protocol; patients will complete 12 sessions of virtual reality exercise application-Nintendo Wii Fit Plus 30-minute training sessions with strengthening exercises for the lower extremities and upper extremities, aerobic and balance exercises. They will do 5 minutes warm-up exercises before the session and 5 minutes cool-down exercises as well as breathing exercises at the end of the session and will participate in a 50-minute treatment session in total.

In the control group treatment protocol, patients will follow the 30-minute video exercise practices for the lower and upper extremities that are similar to Nintendo Wii Fit exercises for the control group at home two days a week. exercises will complete the 50-minute training session. Apart from exercise sessions, patients will record their activities (walking, cycling, swimming…) in daily life forms with their own pedometers. Thus, changes in physical activity levels will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years of age
* to be chronic kidney disease,
* to have chronic kidney disease at least 6 months
* to have no visual hearing impairment

Exclusion Criteria:

* Attending another exercise program,
* to have severe infection (sepsis, peritonitis)
* Having anorexia or other growth retardation,
* Mental retardation,
* Inadequate communication in Turkish,
* Failure to communicate,
* Cardiomyopathy,
* presence of angina pectoris,
* Standing and walking obstacle
* Presence of orthopedic problem
* Cerebrovascular disease
* Patients with lower limb amputation and not using orthosis-prosthesis,
* patients with metastatic carcinoma will not be included in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 Weeks
  The strength of the lower and upper extremity muscles is measured with a digital dynamometer.
Functional Capacity-6-Minute Walking Test | 6 Weeks
  Functional capacity is assessed by 6 minute walk test at the baseline and after 6 weeks

SECONDARY OUTCOMES:
Fatigue | 6 Weeks
  The fatigue parameter is evaluated with the Pediatric Quality of Life Inventory Version 4.0 General Scales (PedsQL), a tool developed specifically to assess the physical, school, emotional, and social domains of health-related quality of life in children previously confirmed in healthy and patient populations. From the physical area of PedsQL individual elements of low energy level will be extracted from both child and parent questionnaires to assess the prevalence of fatigue. The frequency of low energy over the past month is classified as one of four categories: "never"; "hardly"; "sometimes"; "Often / almost always". Overall PedsQL scores, from 0 to 100, higher scores mean better quality of life. PedsQL is scored from the "low energy" item from both parents and child surveys.
Quality of life MEASURE | 6 Weeks
  PedsQLTM 4.0 Quality of Life Scale for Children is used to assess the quality of life of children. PedsQLTM 4.0, with a child / adolescent report and primary caregiver report, is a modular approach to measuring health-related quality of life in healthy children and adolescents in confirmed acute and chronic health conditions in Brazil. The questionnaire evaluates four scales (physical, emotional, social and school functioning) in 23 questions using age-specific forms. Self-report forms are available for children / adolescents aged 5-7, 8-12 or 13-18. Parental reports are available for children aged 2-4, 5-7, 8-12 or 13-18. The questionnaire score ranges from zero to 100 on each scale, and higher values are interpreted to indicate a better quality of life.
Lung Parameters- Forced vital capacity (FVC), forced expiratory volume 1 second | 6 Weeks
  Lung Parameters are measured after 3 repetitive treatments performed by using a digital treatment.
Participation | 6 Weeks
  Participation in the activity is assessed by Scope questionnaire.The Short Child Roller activities and tasks profile (SCOPE) test is a children-specific assessment test. SCOPE is a test that can be used in the age range from birth to 21 years, which evaluates activity participation as person-centered. SCOPE allows the assessment of participation with comparable objective data within the physical, mental and social disabilities of the child. This questionnaire consists of 25 questions and includes 4 questions from the areas of will, habits, interaction and communication skills, processing skills and motor skill activity performance, and 5 questions for the latest environment. High scores indicate good results.
  Children's participation in the activity and their level of entertainment depending on the activity; Short Child Roles Activities and Tasks Profile SCOPE Will and Habits are evaluated by comparing the scores of performance titles before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University of Health Sciences Kanuni Sultan Süleyman Training and research Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No